CLINICAL TRIAL: NCT04223687
Title: Randomized Controlled Trial Evaluating the Impact of Warnings on Sugar-Sweetened Beverages
Brief Title: Impact of Warnings on Sugar-Sweetened Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Robert Wood Johnson Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-0277b; RWJF76290 (Other Grant/Funding Number: Robert Wood Johnson Foundation); K01HL147713 (NIH)
Record Dates: First submitted 2019-12-10; First posted 2020-01-10 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Dietary Habits
Keywords: Food and beverage purchases; Sugar-sweetened beverages; Beverages
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugar-Sweetened Beverage Warning Label (Experimental)
  Interventions: Other: Sugar-Sweetened Beverage Warning Label
- Neutral label (Other)
  Interventions: Other: Neutral label

INTERVENTIONS:
Other: Sugar-Sweetened Beverage Warning Label — Labels with a pictorial warning will be applied to the front-of-package of all sugar-sweetened beverage containers in the mock store. Investigators developed the text and design of these labels based on previous research.
  Arms: Sugar-Sweetened Beverage Warning Label
Other: Neutral label — Neutral labels will be applied to the front-of-package of all sugar-sweetened beverage containers in the mock store. Investigators developed the design of these labels.
  Arms: Neutral label

SUMMARY:
The purpose of this randomized controlled trial is to determine whether pictorial warnings on sugar-sweetened beverages are more effective than neutral labels at reducing parents' purchases of sugar-sweetened beverages for their children. Participants will be parents or guardians of at least one child age 2-12. The trial will take place in a mock convenience store. Participants will be randomly assigned to a pictorial warnings arm in which all sugar-sweetened beverages in the store are labeled with pictorial warnings, or to a control arm in which all sugar-sweetened beverages in the store are labeled with a neutral label. All participants will visit the mock convenience store setup based on their randomized trial arm and be instructed to engage in a shopping task. Participants will complete a computer survey after the shopping task.

DETAILED DESCRIPTION:
Childhood obesity is a major public health problem in the US among racial and ethnic minorities, including among the US's growing Latino population. One promising but understudied policy for addressing childhood obesity is requiring pictorial warnings on the front of sugar-sweetened beverage containers. The impact of pictorial warnings in real-world food retail environments on parents' sugar-sweetened beverage purchasing behavior for their children is unknown. This study will assess the impact of pictorial warnings on parents' sugar-sweetened beverage purchases for their children in a real-world randomized controlled trial. The investigators focus on parents as they are the primary decision-makers and purchasers of food products for children and exert strong influence over their children's dietary intake and food attitudes. Half of participants will be Latino as childhood obesity is a major public health problem among the US's growing Latino population.

Setting: The trial will take place in a mock convenience store setting created for researchers to examine how store and product characteristics influence consumer purchases in a controlled but realistic environment. The store reflects a convenience store's characteristics, with foods, beverages, and household items set at real-world prices.

Recruitment: Participants will be recruited locally via methods including community subject pools, printed flyers posted, and online listings. Interested potential participants will complete a screening questionnaire online, in person, or over the phone to determine their eligibility. If eligible, they will be invited to schedule a time to visit the mock store for the trial.

Informed Consent: At the beginning of the in-person study visit, study staff will explain the consent form. The study staff will ask the participant if he or she has any questions; once the participant consents to the study, both parties will sign the consent form and the participant will receive a copy of the consent form.

Randomization: After the participant signs the consent form, study staff will randomly assign participants to one of the two study arms. Randomization order will be determined a priori. Participants will have an equal chance of being randomized to either arm of the trial.

Assessment: Using an established protocol, participants will visit the mock study convenience store and be given a shopping task to select 1 beverage and 1 snack to purchase for their child ages 2-12. If the participant has more than one child age 2-12, the investigators will randomly select the child they should shop for. At check-out, study staff will record the products selected. Participants will then complete 1 computer-based survey immediately after completing the shopping task. The visit will take approximately 45-60 minutes. At the end of the study, participants will receive an informational handout about sugar-sweetened beverages and healthier alternatives.

Detailed description of the trial arms: Participants will be assigned to either a pictorial warnings arm or a control arm. In the pictorial warnings arm, all sugar-sweetened beverage products in the mock store will be labeled with a pictorial warning label (two different warning labels will be displayed at the same time, but only 1 warning label per product). Investigators developed the text and design of these warning labels using a pre-test. In the control arm, all sugar-sweetened beverage products will be labeled with a neutral label, also developed by the investigators. In both arms, labels will be adhered directly on the front-of-package of sugar-sweetened beverage containers.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Be able to read and speak English or Spanish
* Be able to take a computer survey in English or Spanish
* Be the parent or guardian to at least one child between the ages of 2 and 12 who consumed at least one sugar-sweetened beverage in the week prior to taking the screener

Exclusion Criteria:

* Cannot have participated in the investigator's previous study at the convenience store in the past year
* Cannot live in the same household as another enrolled study participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa G. Hall, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Lindsey S. Taillie, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall MG, Grummon AH, Higgins ICA, Lazard AJ, Prestemon CE, Avendano-Galdamez MI, Taillie LS. The impact of pictorial health warnings on purchases of sugary drinks for children: A randomized controlled trial. PLoS Med. 2022 Feb 1;19(2):e1003885. doi: 10.1371/journal.pmed.1003885. eCollection 2022 Feb. PMID 35104297

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Started | 163 | 163
Completed | 162 | 163
Not Completed | 1 | 0
Not completed — Missing primary outcome | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label | Total
Number analyzed (Participants) | 162 | 163 | 325
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 24 | 21 | 45
  30-39 | 65 | 74 | 139
  40-49 | 53 | 54 | 107
  50+ | 20 | 14 | 34
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 41 | 32 | 73
  Woman | 120 | 130 | 250
  Another gender identity | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Reporting of race/ethnicity was optional. All data collected are included.
  Participants
    Non-Hispanic white | 72 | 70 | 142
    Hispanic white | 9 | 10 | 19
    Hispanic, no race reported | 14 | 15 | 29
    Hispanic, other race(s) | 8 | 9 | 17
    Non-Hispanic Black or African American | 46 | 34 | 80
    Non-Hispanic Asian | 6 | 7 | 13
    Non-Hispanic, more than one race | 3 | 13 | 16
    Non-Hispanic, other race | 0 | 2 | 2
    Data Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 162 | 163 | 325
Time of participation [Count of Participants; unit: Participants] — Time of participation in study, either before the COVID-19 pandemic or during the COVID-19 pandemic.
  Participants
    Pre-pandemic | 64 | 65 | 129
    During pandemic | 98 | 98 | 196

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Purchase at Least 1 Sugar-sweetened Beverage for Their Child
Description: The primary outcome is the percent of participants who selected at least one sugar-sweetened beverage for their child during the shopping task. Purchases will be recorded by the experimenter when they complete the shopping task.
Time Frame: At completion of ~10 minute shopping task, during 1-time study visit
Measure: Number; unit: percentage of participants
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 162 | 163
percentage of participants | 45 | 28
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p < 0.01, Chi-squared — a priori threshold for statistical significance, p<0.05

2. Secondary Outcome: Mean Total Calories Purchased From Sugar-sweetened Beverages
Description: Total calories purchased from sugar-sweetened beverages is defined as the total number of calories of sugar-sweetened beverages in the participant's basket when they complete the shopping task.
Time Frame: At completion of ~10 minute shopping task, during 1-time study visit
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 162 | 163
calories | 82.1 (97.22) | 51.72 (86.82)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p < 0.01, t-test, 2 sided — a priori threshold for statistical significance, p<0.05

3. Secondary Outcome: Mean Intention to Give Sugar-sweetened Beverages to Child
Description: Intention to give sugar-sweetened beverages to child will be measured at post-test by survey. Response options are on a 1 to 7 scale, with higher scores representing a higher intention to give sugar-sweetened beverages to the participant's child.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 160 | 160
score on a scale | 1.85 (0.8) | 1.65 (0.6)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

4. Secondary Outcome: Percentage of Participants Who Noticed Trial Label
Description: Percent of participants who noticed the trial labels will be measured at post-test by survey.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Number; unit: percentage of participants
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 161 | 161
percentage of participants | 47 | 52
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p = 0.37, Chi-squared — a priori threshold for statistical significance, p<0.05

5. Secondary Outcome: Mean Thinking About Harms of Drinking Sugar-sweetened Beverages
Description: How much the participant reports thinking about the health problems caused by drinking sugar-sweetened beverages will be measured at post-test by survey. Response options are on a 1 to 5 scale, with higher scores representing a higher amount of thinking about harms of drinking sugar-sweetened beverages.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 161 | 161
score on a scale | 1.90 (1.25) | 4.21 (0.95)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

6. Secondary Outcome: Mean Negative Affective Reactions
Description: Negative affect will be measured at post-test by survey. Response options are on a 1 to 5 scale, with higher scores representing a higher negative affect reaction.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 160 | 160
score on a scale | 1.51 (0.82) | 3.38 (1.12)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

7. Secondary Outcome: Mean Anticipated Social Interactions
Description: Anticipated social interactions about the study labels will be measured at post-test by survey. Response options are on a 1 to 5 scale, with higher scores representing a higher likelihood of discussing the study labels with others.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 161 | 161
score on a scale | 2.16 (1.32) | 3.89 (1.24)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

8. Secondary Outcome: Percentage of Participants Who Felt More in Control of Healthy Eating Decisions
Description: Percent of participants indicating they felt more in control of healthy eating decisions will be measured at post-test by survey.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Number; unit: percentage of participants
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 161 | 161
percentage of participants | 30 | 73
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p < 0.001, Chi-squared — a priori threshold for statistical significance, p<0.05

9. Secondary Outcome: Mean Perceived Amount of Added Sugar in Sugar-sweetened Beverages
Description: Perceptions of added sugar content in sugar-sweetened beverages will be measured at post-test by survey. Response options are on a 1 to 5 scale, with higher scores representing a higher perceived amount of added sugar in sugar-sweetened beverages.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 160 | 161
score on a scale | 3.99 (0.67) | 4.08 (0.77)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

10. Secondary Outcome: Mean Perceived Likelihood of Child Experiencing Health Problems Due to Sugar-sweetened Beverages
Description: Perceived likelihood of child experiencing sugar-sweetened beverage related health outcomes will be measured at post-test by survey. Response options are on a 1 to 7 scale, with higher scores representing a higher perceived likelihood of child experiencing health problems due to sugar-sweetened beverages.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 152 | 157
score on a scale | 3.95 (0.99) | 4.07 (0.92)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

11. Secondary Outcome: Mean Healthfulness of Sugar-sweetened Beverages for Child
Description: Parents' perceptions about sugar-sweetened beverages' healthfulness for their child will be measured at post-test by survey. Response options are on a 1 to 7 scale, with higher scores representing a higher perceived healthfulness of sugar-sweetened beverages for their child.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 161 | 160
score on a scale | 2.24 (0.80) | 1.98 (0.82)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

12. Secondary Outcome: Mean Appeal of Sugar-sweetened Beverages for Child
Description: Parents' perceptions about sugar-sweetened beverages appeal for their child will be measured at post-test by survey. Response options are on a 1 to 7 scale, with higher scores representing a higher perceived appeal of sugar-sweetened beverages for their child.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 161 | 161
score on a scale | 3.32 (0.96) | 3.24 (0.98)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p = 0.42, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

13. Secondary Outcome: Mean Tastiness of Sugar-sweetened Beverages for Child
Description: Parents' perceptions of tastiness of sugar-sweetened beverages for their child will be measured at post-test by survey. Response options are on a 1 to 7 scale, with higher scores representing a higher perceived tastiness of sugar-sweetened beverages for their child.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 160 | 161
score on a scale | 3.47 (0.89) | 3.30 (0.95)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

14. Secondary Outcome: Mean Injunctive Norms About Limiting Child's Sugar-sweetened Beverages
Description: Injunctive norms about limiting child's sugar-sweetened beverage consumption will be measured at post-test by survey. Injunctive norms refer to perceived approval from people important in the participant's life. Response options are on a 1 to 5 scale, with higher scores representing higher perceived approval about limiting their child's sugar-sweetened beverages.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 158 | 158
score on a scale | 3.21 (1.33) | 3.60 (1.20)
Statistical Analysis 1: Comparison: Neutral Label vs Sugar-Sweetened Beverage Warning Label; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney) — a priori threshold for statistical significance, p<0.05

15. Other Pre Specified Outcome: Mean Anticipated Avoidance of Label
Description: Avoidance of the study labels will be measured at post-test by survey. Response options are on a 1 to 5 scale, with higher scores representing a higher amount of avoidance of looking at the study labels.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 160 | 161
score on a scale | 1.94 (1.2) | 3.43 (1.3)

16. Other Pre Specified Outcome: Mean Perceived Message Effectiveness
Description: Perceived message effectiveness of the study labels will be measured at post-test by survey. Response options are on a 1 to 5 scale, with higher scores representing a higher perceived message effectiveness of the study labels.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 159 | 153
score on a scale | 2.0 (1.3) | 4.2 (.9)

17. Other Pre Specified Outcome: Mean Policy Support
Description: Support for sugar-sweetened beverage health warning labels will be measured at post-test by survey. Response options are on a 1 to 4 scale, with higher scores representing a higher amount of support for a sugar-sweetened beverage health warning label policy.
Time Frame: Post-test computer survey within 30 minutes following completion of ~10 minute shopping task
Population: Assessed for people who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neutral Label | Sugar-Sweetened Beverage Warning Label
Number analyzed (Participants) | 161 | 161
score on a scale | 3.00 (0.9) | 3.49 (0.8)

ADVERSE EVENTS:
Time Frame: From the time of signing the Informed Consent through study completion, an approximate total of up to 1 hour.
Arm/Group | Sugar-Sweetened Beverage Warning Label | Neutral Label
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/163
Other Adverse Events (participants affected / at risk) | 0/163 | 0/163

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT04223687/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT04223687/SAP_000.pdf